CLINICAL TRIAL: NCT00251485
Title: A Phase II Trial of Modified FOLFOX 6 and Cetuximab in First Line Treatment of Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Veeda Oncology (Other)
Collaborators: Bristol-Myers Squibb (Industry); Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-03-002
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Colorectal Cancer
Keywords: Metastatic 1st line colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cetuximab — Cycle 1: 400 mg/m2 (given as a 2-hour infusion) on Day 1, then 250 mg/m2, Day 8 (given as a 1-hour infusion) subsequent cycles:250 mg/m2, Day 1 and Day 8 (given as a 1-hour infusion)

SUMMARY:
This is a Phase II, open label, non-randomized study in patients with histologically or pathologically confirmed diagnosis of stage IIIB/IV, EGFR+ adenocarcinoma of the colon or rectum who have not received prior chemotherapy for their metastatic disease.

Primary Study Endpoint:

To assess the response rate, progression-free survival, and overall safety profile of a modified FOLFOX 6 plus cetuximab regimen in the first-line treatment of patients with metastatic colorectal cancer.

Secondary Study Endpoint(s):

To assess overall survival of patients with metastatic colorectal cancer who receive first-line therapy with a modified FOLFOX 6 + cetuximab regimen.

DETAILED DESCRIPTION:
The current treatment options for metastatic colon cancer are in need of further improvement. The three-drug combination of oxaliplatin with 5-FU/LV for the first-line treatment of metastatic colorectal cancer has shown a significant increase in response rate compared to IFL (irinotecan and bolus 5-FU plus leucovorin ) and IROX (irinotecan plus oxaliplatin. Cetuximab has shown activity with and without irinotecan in subjects with colorectal cancer refractory to irinotecan alone.30,31 Cetuximab has also been shown to be safe and effective when administered with infusional 5-FU/folinic acid plus irinotecan. These results suggest that the addition of cetuximab to a 5-FU/LV/oxaliplatin-based regimen (FOLFOX) used in the 1st line setting may lead to the development of more treatment options for subjects with advanced colorectal cancer.

This is a Phase II, open label, non-randomized study in patients with histologically or pathologically confirmed diagnosis of stage IIIB/IV, EGFR+ adenocarcinoma of the colon or rectum who have not received prior chemotherapy for their metastatic disease.

Patients will receive a modified FOLFOX 6 regimen (5-FU, leucovorin, and oxaliplatin) every 2 weeks in combination with cetuximab given weekly.

Patients will be evaluated for response and progression-free survival. Overall survival will also be evaluated, as well as the safety profile of the regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have signed an IRB approved informed consent.
2. Patients with histologically or pathologically documented, stage IIIB or IV adenocarcinoma of the colon or rectum.
3. Patients with disease that is not amenable to potentially curative resection (i.e., inoperable metastatic disease).
4. Patients with tumors that are EGFR + by IHC staining.
5. Patients with ECOG Performance status of 0 or 1.
6. Patients, 18 years and older, must either be not of child bearing potential or have a negative serum pregnancy test within 7 days prior to registration. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or they are postmenopausal.
7. Bone marrow function: absolute neutrophil count (ANC) > or = 1,500/uL, equivalent to Common Terminology Criteria for Adverse Events (CTCAE, version 3) Grade 1. Platelets > or = 100,000/uL (CTCAE Grade 0 - 1).
8. Renal function: creatinine < or = 1.5 x institutional upper limit of normal (ULN), CTCAE Grade 1.
9. Hepatic function: bilirubin < or = 1.5 x ULN, CTCAE Grade 1. AST < or = 2.5 x ULN, CTCAE Grade 1.

Exclusion Criteria:

1. Patients who received prior chemotherapy for metastatic disease. Prior adjuvant therapy with 5FU/LV and/or irinotecan is allowed provided it was completed at least 6 months prior to enrollment in this study.
2. Patents who received prior oxaliplatin.
3. Patients who received prior cetuximab or other therapy which specifically and directly targets the EGF pathway.
4. Patients with acute hepatitis.
5. Patients with active or uncontrolled infection.
6. Patients with a significant history of cardiac disease, i.e., uncontrolled hypertension, unstable angina, and congestive heart failure.
7. Prior allergic reaction to chimerized or murine monoclonal antibody therapy.
8. Any concurrent chemotherapy not indicated in the study protocol or any other investigational agent.
9. Patients with peripheral neuropathy > grade 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2004-03; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
To assess the response rate, progression-free survival, and overall safety profile of a modified FOLFOX 6 plus cetuximab regimen in the first-line treatment of patients with metastatic colorectal cancer. | unk

SECONDARY OUTCOMES:
To assess overall survival of patients with metastatic colorectal cancer who receive first-line therapy with a modified FOLFOX 6 + cetuximab regimen | unk

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Boccia, MD, Principal Investigator — Veeda Oncology
Locations (1):
- Veeda Oncology, Houston, Texas, United States